CLINICAL TRIAL: NCT05974592
Title: The Effect of Nurse-Led Diabetic Foot Self-Management Training Program on Diabetic Foot Knowledge, Foot Care Behavior, and Self-Efficacy Levels in Patients With Type 2 Diabetes Mellitus: A Randomized Controlled Study
Brief Title: The Effect of Nurse-Led Diabetic Foot Self-Management Training Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Emine Celik Polat, Nurse, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 145/10
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Foot
Keywords: diabetic foot; Patient Education; Foot Care; Self-Efficacy; Nurse
MeSH Terms: conditions — Diabetic Foot | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): To the participants in the intervention group; the "Diabetic Foot Self-Management Training Program (DFSMTP)" will be implemented. Printed, visual, and audio training materials will be used within this training program's scope. Training will be held in the Diabetes Education Room in line with the content of DFSMTP prepared by the researcher after determining the appropriate day and time with the participants. Written (training booklet) and visual (computer and PowerPoint presentation) training materials will be used during this training. The printed training booklet will be delivered to the participants at the end of the training. DFSMTP will be held in three sessions on the same day. In order to reinforce the learning of the participants in the intervention group, DFSMTP will also be video recorded with the presentation of the researcher and this recording will be transferred to the DFSMTP YouTube channel to be created by the researcher.
  Interventions: Other: Education
- Control Group (No Intervention): To the participants in the control group; General information about the anatomy and physiology of the pancreas will be explained with the verbal lecture technique. Participants in this group will receive the training only once. Following the completion of the research, the printed training booklet and YouTube channel link information will be shared with the participants.

INTERVENTIONS:
Other: Education — Diabetic Foot Self-Management Training Program will be implemented.
  Arms: Intervention Group

SUMMARY:
Diabetic foot is one of the most important chronic complications of Diabetes Mellitus (DM), which is a global health problem today. Diabetic foot not only affects the individual's quality of life, body image, role performance, and social and economic structure of the family and society but also creates a serious burden on the individual's family and health system. Therefore, some approaches that include foot and nail care, shoe and sock(s) selection, nutrition, and exercise practices are recommended to prevent diabetic foot and to increase functional capacity, without the need for surgical treatment. It is crucial to maintain these recommended approaches throughout the patient's life to ensure effective management of the diabetic foot. This study aims to determine the effect of the nurse-led diabetic foot self-management training program on diabetic foot knowledge, foot care behavior, and self-efficacy level in patients with type 2 DM. This study was planned in a randomized controlled design. The population of the study will consist of type 2 DM patients who do not use insulin therapy and who applied to University of Health Sciences Diskapi Yildirim Beyazit Training and Research Hospital Diabetes outpatient clinic and Diabetes Education outpatient clinic between September 2022 and September 2023. According to the power analysis, 38 participants are targeted to be reached in total. Data will be collected with a Personal Information Form, Diabetic Foot Information Scale, Foot Care Behavior Scale, Diabetic Foot Care Self-Efficacy Scale, and Diabetic Foot Evaluation Form. As a result of this study, it is expected that the nurse-led diabetic foot self-management training program will increase the diabetic foot knowledge, foot care behavior and self-efficacy levels of diabetic foot knowledge, foot care behavior, and self-efficacy level in patients with type 2 DM.

DETAILED DESCRIPTION:
The data to be obtained from the research will be evaluated by transferring them to the IBM SPSS (Statistical Packages for the Social Sciences) Statistics 23 program. Descriptive statistics for continuous variables (mean, standard deviation, median, minimum, maximum), frequency distribution will be used for categorical variables. Differences between categorical variables will be evaluated with Chi-square test and Fisher Exact test, and relations between numerical variables will be evaluated with Spearman Correlation Analysis. The conformity of the data to the normal distribution will be evaluated with the Shapiro Wilk test of normality and Q-Q graphs. Accordingly, if the parametric test assumptions are met, the Significance Test of the Difference Between Two Means in the comparison of independent group differences; If the parametric test assumptions cannot be met, the Mann-Whitney U test will be used. In dependent group comparisons, if parametric test assumptions are met, Analysis of Variance in Repeated Measurements and Significance Test of Difference Between Two Spouses; Friedman Test and Wilcoxon Paired Two Sample Test will be used when parametric test assumptions are not met. A value of p ≤ 0.05 will be considered statistically significant in all analyses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Having Type 2 DM for 1 year or more,
* HbA1C level of 7.5% and below,
* Not using insulin therapy,
* Able to use WhatsApp himself or his relatives
* Individuals who volunteer to participate in the research will be included in the research.

Exclusion Criteria:

* Pregnant or having a pregnancy plan,
* Mental or cognitive impairment
* Having a diabetic foot diagnosis confirmed by a physician,
* Individuals with advanced complications (retinopathy, nephropathy, peripheral arterial disease, etc.) associated with DM diagnosed by a physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Diabetic Foot Care Self-Efficacy Scale (DABS) | It will be applied to the participants at baseline, pre- training, as well as at the 1 month and 8 month follow ups.
  It is a Likert-type scale developed by Quarles in 2005 in accordance with western culture to determine the self-perception of diabetic patients in performing diabetic foot care activities. Self-efficacy is measured by scoring between 0 and 10. The scale consists of 9 items. The 9 statements that make up the scale are evaluated on the 11-digit visual scale, which is stated as "I'm not sure = 0 and very sure = 10". The lowest score of the scale is 0, and the highest score is 90. As the score obtained from the scale increases, the diabetic foot self-efficacy level increases. The Cronbach's alpha value of the sub-dimensions of the scale was 0.94. The validity and reliability study of the scale in the Turkish population was carried out by Kir Bicer and Enc (2014), and the Cronbach alpha value was found to be 0.86.
Diabetic Foot Knowledge Scale (DABI) | It will be applied to the participants at baseline, pre- training, as well as at the 1 month and 8 month follow ups.
  The Turkish validity-reliability study of the scale developed by Alexandra et al.(2001) to evaluate the diabetic foot information of diabetic patients was conducted by Biçer and Enç (2011). The scale consists of 5 items. Diabetic foot knowledge is evaluated using a 5-item DABÖ, a subscale. The Cronbach alpha value of the Turkish version of the scale was 0.58.
Foot Care Behavior Scale (USAS) | It will be applied to the participants at baseline, pre- training, as well as at the 1 month and 8 month follow ups.
  There are 16 items in the scale developed by Borges (2007) in line with the criteria of the American Diabetes Association (ADA) in order to improve foot care behaviors in patients with diabetes (51). The Turkish validity and reliability study was conducted by Kır Biçer and Enç (2014), and it was adapted as a 15-item Foot Care Behavior Scale in line with expert opinions. Each item in the scale is rated on a Likert-type scale between 1 (never) and 5 (always do). The lowest score that can be obtained from the scale is 15; the highest score is 75; High scores indicate that foot care behavior is sufficient. The Cronbach's alpha value for the Turkish version of the scale was found to be 0.83 (high reliability).

SECONDARY OUTCOMES:
Diabetic Foot Evaluation Form (DADF) | It will be applied to the participants at baseline, pre- training, as well as at the 1 month and 8 month follow ups.
  Physical examination of the foot will be done by the thesis student using the Diabetic Foot Evaluation Form developed by the Diabetes Nursing Association Diabetic Foot Study Group. In this form, the fingertips, foot body and leg heat, humidity, presence of edema; nail cutting, deformity, finger examination, presence of dorsalis pedis and tibialis posterior pulses, foot sensation test, muscle strength, ankle-arm index, deformities and shoes and ulcer evaluation if any.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No